CLINICAL TRIAL: NCT05285254
Title: The Impact of the Certified Child Life Specialist in the Pediatric Primary Care Clinic on Children's Pain During Routine Immunizations
Brief Title: The Impact of the Certified Child Life Specialist on Children's Pain During Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Seth W. Gregory, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-002328
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunization Administration with Certified Child Life Specialist Support (CCLS) (Experimental): Nursing will administer immunizations to children with the support of a CCLS
  Interventions: Other: Certified Child Life Specialist Support
- Current Standard of Care for Immunization Administration (No Intervention): Nursing will administer immunizations to children per their current standard of care.

INTERVENTIONS:
Other: Certified Child Life Specialist Support — Provides psychosocial care to children and families confronting stressful and painful situations
  Arms: Immunization Administration with Certified Child Life Specialist Support (CCLS)

SUMMARY:
The purpose of this study is to provide the first systematic evidence that Certified Child Life Specialists reduce pain during vaccine administration and improve caregiver visit satisfaction in the pediatric primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-12 years of age presenting to MCHS Red Wing for a well child examination and vaccine administration.
* Parents or caregivers of any age presenting to well child examination with child.
* Legal guardians of all participants must provide verbal consent.
* Patients must provide verbal assent for participation.Verbal assent will be waived for children younger than 6 years.

Exclusion Criteria:

* Children with autism or other severe developmental disabilities.
* Children must be able to communicate pain before and after vaccine administration using the FPS-R.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported pain | Post vaccine administration, approximately 1 hour
  Measured using the Faces Pain Scale-Revised (FPS-R). This is a self-report measure of pain validated for children ages 4-16 years of age and approved for the assessment of pediatric pain at Mayo Clinic. The scale utilizes different faces to score the sensation of pain on a 0-to-10 metric.
Observed Negative Emotional Responses | Post vaccine administration, approximately 1 hour
  Measured using the Children's Emotional Manifestation Scale (CEMS). The CEMS consists of five categories (facial expression, vocalization, activity, interaction, and level of cooperation) with each category scored from 1 to 5, with summed scores from 5 to 25. Higher scores represent more negative emotional behaviors. The scale was initially validated for children 7-12 years of age but has been subsequently used by other studies for children as young as 4 years of age.

SECONDARY OUTCOMES:
Caregiver visit satisfaction | Post vaccine administration, approximately 1 hour
  Measured by a caregiver satisfaction survey. This is a self-report 6-item survey to rate satisfaction level during child's immunization on a scale of 1=very satisfied and 5=dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Gregory, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Red Wing, Red Wing, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials